CLINICAL TRIAL: NCT01065467
Title: A Pilot/Phase I Study of Panobinostat (LBH589) in Patients With Metastatic Melanoma
Brief Title: Panobinostat (LBH589) in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Novartis (Industry)
Responsible Party: Principal Investigator, F. Stephen Hodi, MD, Melanoma Disease Center Director, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-427; CLBH589BUS64T (Other: Novartis)
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Melanoma; Malignant Melanoma
Keywords: LBH589; panobinostat
MeSH Terms: conditions — Melanoma | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): LBH589
  Interventions: Drug: LBH589

INTERVENTIONS:
Drug: LBH589 — Taken orally three times per week.
  Other Names: Panobinostat

SUMMARY:
The purpose of this research study is to determine the safety of LBH589 as well as to find out what side effects it may cause and how effective it is against melanoma. LBH589 is a drug which may slow down the growth of cancer cells or kill cancer cells by blocking certain enzymes, which are proteins normally produced by cells. These enzymes are known to play an important role in the development and reproduction of cancer cells. It is believed that LBH589 works by helping to promote the activity of enzymes which turn on the mechanisms in our cells that suppress cells from becoming cancerous.

DETAILED DESCRIPTION:
* Each treatment cycle lasts 28 days. During the cycles, participants will be taking LBH589 three days a week(Monday, Wednesday and Friday) every other week.
* During all treatment cycles participants will have a physical exam and will be asked general questions about their health and specific questions about any problems that they may be having. Participants will be seen at least weekly during the first cycle and then at least monthly while they remain on the study.
* Blood tests will be taken to check blood cell counts, how well their organs are functioning and to test for any infections. These blood samples will be obtained prior to the start of every cycle and at least weekly during the first cycle on this study.
* If the participant is a woman of child-bearing potential, she will be asked to undergo either a blood test or provide a urine specimen to check for pregnancy before starting cycle 1 and prior to the start of all subsequent cycles.
* As it is possible for LBH589 to affect the rhythm of the heart, EKGs will be checked frequently during participation on this study. These EKGs will be performed at the following time points: Cycle 1, day 1; Cycle 1, day 5; Cycle 1, Day 8; Cycle 1 day 15; and day 1 of each subsequent cycles.
* CT scans of the chest, abdomen and pelvis and an MRI of the brain will be performed after every 2 cycles or every 56 days.
* A second sample of the participant's tumor will be removed at the end of the first cycle on study.
* Participants will be in this research study for at least 2 months and may continue on the study of they are benefitting from the drug and are not experiencing any serious side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic melanoma
* Measurable disease
* 18 years of age or older
* ECOG performance status of 0, 1 or 2
* Normal organ and marrow function as outlined in the protocol
* Women of childbearing potential must have a negative serum pregnancy test within 7 days of the first administration of study treatment and must be willing to use two methods of contraception during the study and for 3 months after last study drug administration
* Clinically euthyroid
* Biopsiable disease: Disease must be in the opinion of the treating investigator biopsiable such that there are minimal risks involved

Exclusion Criteria:

* Chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* May not be receiving any other study agents, anti-cancer therapy or radiation therapy
* Known brain metastases or any history of brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to LBH589
* Concomitant use of drugs with a risk of causing torsades de pointes
* Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer
* Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first LBH589 treatment
* Impaired cardiac function
* Uncontrolled hypertension
* Patients with unresolved diarrhea grade 2 or greater
* Impairment of the gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral LBH589
* Pregnant or breastfeeding women
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy; individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Patients with known positivity for human immunodeficiency virus (HIV) or hepatitis C
* Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent
* Uncontrolled and/or severe intercurrent illness including, but not limited to ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2017-03-13 (Actual)

PRIMARY OUTCOMES:
To obtain an early evaluation of efficacy by response rate using RECIST criteria. | 2 years

SECONDARY OUTCOMES:
Tp determine whether LBH589 effectively down regulates MITF in biopsy specimens of treated metastatic melanoma patients | 2 years
To estimate the disease control rate using RECIST criteria | 2 years
To estimate time to disease progression. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: F. Stephen Hodi, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States